CLINICAL TRIAL: NCT02724241
Title: The Effects of Electronic Cigarettes on Sympathetic Nerve Activity and Oxidative Stress
Brief Title: E-Cigarettes and SNA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Los Angeles (Other)
Responsible Party: Principal Investigator, Holly R Middlekauff, Professor of Medicine, University of California, Los Angeles
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: 14-000731
Record Dates: First submitted 2016-03-17; First posted 2016-03-31 (Estimated); Last update posted 2021-12-20 (Actual); Status verified 2021-12

CONDITIONS: Nicotine Dependence
Keywords: nicotine; autonomic tone; oxidative stress
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Nicotine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- nicotine (Experimental): use of an e-cigarette filled with liquid with nicotine
  Interventions: Other: one time exposure to e-cig with nicotine
- no nicotine (Experimental): Use of an e-cigarette filled with liquid without nicotine
  Interventions: Other: One time exposure to e-cigarette without nicotine
- sham comparator (Sham Comparator): Use of empty e-cigarette (sham control)
  Interventions: Other: one time exposure to empty e-cigarette

INTERVENTIONS:
Other: one time exposure to e-cig with nicotine — one time exposure to e-cigarette vapor with nicotine
  Arms: nicotine
Other: One time exposure to e-cigarette without nicotine — One time exposure to e-cig without nicotine
  Arms: no nicotine
Other: one time exposure to empty e-cigarette — one time exposure to empty e-cigarette (sham control)
  Other Names: sham control
  Arms: sham comparator

SUMMARY:
Randomized controlled trial of electronic cigarettes with nicotine, without nicotine, and sham control, on sympathetic nerve activity and markers of oxidative stress.

DETAILED DESCRIPTION:
Participants will use an electronic cigarette on 3 occasions: 1) with nicotine, 2) without nicotine, 3) sham control, and measures of autonomic tone, including heart rate variability (HRV) and sympathetic nerve activity (MSNA: microneurography), and oxidative stress will be measured pre and post exposure.

ELIGIBILITY:
Inclusion Criteria:

Healthy

Exclusion Criteria:

* Cardiac disease
* Respiratory disease
* Diabetes mellitus

Ages: 21 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2015-04; Primary Completion 2021-12 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Heart Rate variability | 10 minutes after exposure
  Heart rate variability is a measure of autonomic tone
Paraoxonase | less than 1 hour after exposure
  plasma oxidative stress

SECONDARY OUTCOMES:
muscle sympathetic nerve activity | 10 minutes after exposure
  Muscle sympathetic nerve activity (MSNA)

CONTACTS AND LOCATIONS:
Locations (1):
- UCaliforniaLA, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No